CLINICAL TRIAL: NCT03866603
Title: Rostock International Parkinson's Disease Study: an International, Multicenter, Epidemiological Observational Study
Brief Title: Rostock International Parkinson's Disease Study (ROPAD)
Acronym: ROPAD
Status: Active, not recruiting | Type: Observational
Sponsor: CENTOGENE GmbH Rostock (Industry)
Responsible Party: Sponsor
Other Study IDs: ROPAD 01-2019
Record Dates: First submitted 2019-03-01; First posted 2019-03-07 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Parkinson´s Disease
Keywords: Parkinson´s disease; Biomarker; LRRK2; GBA; PD Genetics
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample applied on the Dry Blood Spot (DBS) Filtercard (Centocard®)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Parkinson´s disease individuals: * The participant has been clinically diagnosed with Parkinson's disease within the last 5 years (≤ 5 years)
  * The participant is between 30 and 80 years old

SUMMARY:
Rostock International Parkinson's Disease Study - An International, multicenter, epidemiological observational study aiming at identification of LRRK2-positive patients, the recruitment of 25,000 PD participants and the establishment of a candidate biomarker in the LRRK2-positive cohort.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is one of the most common neurodegenerative disorders worldwide, affecting approximately 1% of individuals older than 60 years and causes progressive disability.

Clinical signs and symptoms of PD include the following: asymmetric tremor at rest, bradykinesia, muscle rigidity, postural instability, gait abnormalities including festination and freezing. Onset is typically after the age of 50 years and the disease is commonly slowly progressive. The most common initial finding of PD is a resting tremor in the upper extremity. Over time, participants experience progressive bradykinesia, rigidity, and gait difficulty, while the axial posture becomes progressively flexed. Non-motor symptoms are common in all stages of Parkinson disease and they include constipation, seborrhea, hyposmia or anosmia, sympathetic denervation of the heart, depression and/or apathy, sleep disturbances, cognitive decline and dementia. They may appear prior to the movement disorder and can be used as preclinical markers of PD.

PD is mostly considered as idiopathic disease; however more and more data suggest that it is a disease that involves interaction of genetic and environmental factors. The most common monogenic form and the one most closely resembling idiopathic PD is LRRK2 (Leucine-rich repeat kinase 2 gene) associated PD.

The most common monogenic form and the one most closely resembling idiopathic PD is LRRK2 (Leucine-rich repeat kinase 2 gene) associated PD. First identified in 2004, LRRK2 mutations are currently still the most commonly known cause of PD and account for up to ~40% of all Parkinson's disease cases in select populations. The majority of reported LRRK2-positive PD patients are Caucasian (63%), whereas all other ethnicities comprise ~10% or fewer patients of described mutation carriers despite clusters in the Ashkenazi Jewish and Arab Berber populations. With respect to country of origin, the majority of patients were re-ported to reside in Italy or Spain (14% each), Great Britain (10%) or Norway (9%). Definitely pathogenic variants identified in LRRK2 include p.G2019S, p.R1441C/G/H, p.N1437H, p.Y1699C, and, p.I2020T. Of these, the p.R1441G mutation is particularly frequent, as it represents a founder mutation in the Basque population where it is responsible for 46% of all familial PD. Very rarely, this mutation has also been observed in other populations where it arose on a different haplotype. LRRK2 p.Gly2019Ser mutation accounts for about 0.5% simplex cases and >5% familial cases in various ethnic groups worldwide. Furthermore, genome-wide association studies have identified common polymorphisms in LRRK2 that associate with idiopathic PD, implicating LRRK2 function in susceptibility to late-onset PD in individuals without pathogenic mutations.

LRRK2 mutations cause PD with age-related penetrance and clinical features identical to late-onset sporadic PD. Biochemical studies support an increase in LRRK2 kinase activity and a decrease in GTPase activity for kinase domain and Roc-COR mutations, respectively. Strong evidence exists that LRRK2 toxicity is kinase dependent, leading to extensive efforts to identify selective and brain-permeable LRRK2 kinase inhibitors for clinical development. LRRK2 kinase inhibition is currently one of the most prevailing disease-modifying therapeutic strategies for PD. Thus, LRRK2 kinase inhibitors are in development as potential Parkinson's disease therapeutics.

Furthermore, there is now evidence showing that LRRK2 expression and phosphorylation levels have a potential as markers of Parkinson's disease. Recently, the presence of Lrrk2 was confirmed in exosomes from human biofluids, including urine and cerebrospinal fluid. Moreover, elevated LRRK2 autophosphorylation was identified in brain-derived and peripheral exosomes in LRRK2-mutation carriers. In summary, it has been shown that markers of LRRK2 activity and function may be detected in human blood and that they are relevant for pathogenesis if PD.

Thus, the biochemical analyses of human blood from LRRK2 positive participants and LRRK2 negative participants create a strong base for the development of PD-related biomarkers. This biomarker may in turn be even more accessible than genetic testing and it may serve for diagnosis, prognosis, and prediction of PD.

ELIGIBILITY:
* Informed consent is obtained from the participant
* The participant has been clinically diagnosed with Parkinson's disease within the last 5 years (≤ 5 years)
* The participant is between 30 and 80 years old

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants clinically diagnosed with Parkinson's Disease (PD)
Sampling Method: Non-Probability Sample
Enrollment: 25000 (Estimated)
Dates: Start 2019-05-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To investigate the prevalence of genetic etiologies of PD | 79 months

SECONDARY OUTCOMES:
To identify LRRK2-positive PD participants from the primary strata, Establishment of a biomarker in the LRRK2-positive cohort | 79 months

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bauer, MD, Principal Investigator — CENTOGENE GmbH
Locations (110):
- United States (26):
  - Tucson Neuroscience Research, Tucson, Arizona
  - Pharmacology Research Institute, Encino, California
  - Neuro-Pain Medical Center, Fresno, California
  - University of California (UC) San Diego, La Jolla, California
  - Loma Linda University, Loma Linda, California
  - Pharmacology Research Institute, Los Alamitos, California
  - Pharmacology Research Institute, Newport Beach, California
  - Parkinson's Disease and Movement Disorder Center of Baco Raton, Baco Raton, Florida
  - Linfritz Research Institute, Coral Gables, Florida
  - Renstar Medical Research, Ocala, Florida
  - University of South Florida, Tampa, Florida
  - Vero Beach Neurology & Research Institute, Vero Beach, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Northshore University HealthSystem, Evanston, Illinois
  - Indiana University, Department of Neurology, Indianapolis, Indiana
  - Michigan Institute for Neurological Disorders, Farmington Hills, Michigan
  - WR-CRCN, Las Vegas, Nevada
  - Neuroscience Research Institute of NJ, Toms River, New Jersey
  - Dent Neurologic Institue, Amherst, New York
  - Stony Brook University School of Medicine, Brookhaven, New York
  - South Shore Neurologic Associates, Patchogue, New York
  - Duke University, Department of Neurology, Durham, North Carolina
  - M3 Wake Research, Inc., Raleigh, North Carolina
  - WR-ClinSearch, LLC, Chattanooga, Tennessee
  - Booth Gardner Parkinson's Care Center, Kirkland, Washington
  - Inland Northwest Research, Spokane, Washington
- Qendra Spitalore University, Tirana, Albania
- Belgium (4):
  - University Hospital of Antwerp, Antwerp
  - UZ Leuven, Campus Gasthuisberg, Leuven
  - Department of Neurology, Centre Hospitalier Universitaire (CHU) de Leige, Liège
  - AZ Damiaan, Department of Neurology, Ostend
- Brazil (13):
  - Hospital das Clínicas da Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais
  - Hospital Ophir Loyola, Belém, Pará
  - Federal University of Health Science of Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Universidade Metropolitana De Santos, Santos, São Paulo
  - Hospital Universitário Walter Cândido/ Universidade Federal do Ceará, Ceará
  - Hospital Angelina Caron, Curitiba
  - Fundação Hospital Adriano Jorge, Manaus
  - Carolina São Souza, Ribeirão Preto
  - Faculdade de Medicina de Ribeirão Preto - USP, Ribeirão Preto
  - Hospital Universitario Pedro Ernesto (HUPE), Rio de Janeiro
  - Universidade Federal de São Paulo, UNIFESP, São Paulo
  - Clinica de Neurocirurgia E Neurofisiologia Ltda, São Paulo
  - Instituto Israelita de Ensino e Pesquisa Albert Einstein, São Paulo
- Toronto Western Hospital, University Health Network, University of Toronto, Toronto, Ontario, Canada
- Groupe Hospitalier Paris Saint-Joseph, Paris, France
- Germany (18):
  - Universitätsklinik für Neurologie, Aachen
  - Neurologisches Fachkrankenhaus für Bewegungsstörungen / Parkinson, Beelitz
  - Kliniken Beelitz, Beelitz-Heilstätten
  - Charite University Medicine, Berlin
  - Gertrudis-Kliniken im Parkison-Zentrum, Biskirchen
  - St. Josef-Hospital, Bochum
  - Universitätsklinikum Carl Gustav Carus die Dresdner, Dresden
  - Asklepios Klinik Barmbek, Hamburg
  - Universitätsklinik Hamburg-Eppendorf, Hamburg-Eppendorf
  - Universitätsklinik für Neurologie, Jena
  - Paracelsus Elena-Klinik, Kassel
  - Universitätsklinikum Schleswig-Holstein, Klinik für Neurologie, Kiel
  - Universitätsklinikum Leipzig, Leipzig
  - Universitätsklinikum Schleswig-Holstein Campus Lübeck, Lübeck
  - Universitätsklinikum Marburg Klinik und Poliklinik für Neurologie Parkinson Netzwerk Allianz Marburg (PANAMA), Marburg
  - Diakonie-Klinikum Schwäbisch Hall gGmbH, Schwäbisch Hall
  - Asklepios Fachklinikum Stadtroda Klinik für Neurologie, Schmerztherapie und Schlafmedizin, Stadtroda
  - Universitätsklinikum Würzburg, Würzburg
- Mediterraneo Hospital, Athens, Greece
- Israel (10):
  - Samson Assuta Ashdod University Hospital, Ashdod
  - Barzilai Medical Center, Ashkelon
  - Soroka Medical Center, Beersheba
  - Shamir Medical Center, Be’er Ya‘aqov
  - RAMBAM Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Medical Center, Jerusalem
  - Rabin MC, Beilinson Campus, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center - TASMC, Tel Aviv
- Italy (4):
  - AOUP Secondo Policlinico Federico II Napoli, Napoli
  - Università di Pavia, Dipartimento di Medicina Molecolare, Pavia
  - Asmn - Irccs, Reggio Emilia
  - I.R.C.C.S. San Raffaele Pisana, Roma
- St. Olav's Hospital, Trondheim, Norway
- Portugal (2):
  - Neurology Department, Hospital de Santa Maria, Lisbon
  - Centro Hospitalar Universitário de São João, Porto
- Spain (12):
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Clinico Universitario Santiago de Compostela, Santiago de Compostela, Corunna
  - Hospital Universitario de La Princesa, Madrid, Madrid
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital Universitario Fundación Alcorcón, Alcorcón
  - Instituto Investigacion Biocruces, Barakaldo
  - Hospital General Unversitario Gregorio Marañón, Madrid
  - HM CINAC | Integrated Neuroscience Center, Móstoles
  - Clinica Universidad de Navarra (CUN), Pamplona
  - Hospital Universitario Donostia, San Sebastián
  - University Hospital Marqués de Valdecilla, Santander
- Turkey (Türkiye) (4):
  - Cukurova University Faculty of Medicine, Sarıçam, Adana
  - Istanbul Faculty of Medicine, Istanbul, Istanbul
  - Mersin Faculty of Medicine, Mersin, Mersin
  - Koc University Hospital, Istanbul
- United Kingdom (12):
  - Fairfield General Hospital, Bury
  - University of Dundee, Dundee
  - University of Edinburgh, Edinburgh
  - Royal Devon and Exeter Hospital, Exeter
  - Imperial College Healthcare NHS Trust, London
  - Newcastle University, Clinical Ageing Research Unit, Newcastle upon Tyne
  - University of Oxford, Nuffield Department of Clinical Neurosciences, Oxford
  - University of Plymouth, Plymouth
  - Royal Preston Hospital, Department of Neurology, Preston
  - Salford Royal NHS Foundation Trust, Salford
  - Royal Cornwall Hospitals Nhs Trust, Truro
  - Yeovil District Hospital, Yeovil

IPD SHARING:
Plan to Share IPD: No
The plan will be defined at a later stages

REFERENCES:
- [Background] Baumann CR. Epidemiology, diagnosis and differential diagnosis in Parkinson's disease tremor. Parkinsonism Relat Disord. 2012 Jan;18 Suppl 1:S90-2. doi: 10.1016/S1353-8020(11)70029-3. PMID 22166466
- [Derived] Dayan R, Bick AS, Weill C, Bauer M, Erdman HB, Israel Z, Bergman H, Levin N, Arkadir D. Atrophy-related corticospinal changes in advanced Parkinson's disease are associated with the genetic etiology of the disease. J Parkinsons Dis. 2024 Nov;14(8):1584-1593. doi: 10.3233/JPD-240267. Epub 2024 Nov 4. PMID 39957202